CLINICAL TRIAL: NCT05575726
Title: Effects of Neutrophil Extracellular Traps and Damage-associated Molecular Pattern Molecules on Long Term Use of Macrolides in Adults With Chronic Respiratory Disease：A Prospective Observational Study.
Brief Title: Effects of Neutrophil Extracellular Traps and Damage-associated Molecular Pattern Molecules on Long Term Use of Macrolides in Adults With Chronic Respiratory Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-230
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2021-12

CONDITIONS: Chronic Respiratory Disease
Keywords: neutrophil extracellular traps; damage-associated molecular pattern molecules; macrolides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum

SUMMARY:
The purpose of this study is to investigate the effects of neutrophil extracellular traps and damage-associated molecular pattern molecules on long term use of macrolides in adults with chronic respiratory disease.

DETAILED DESCRIPTION:
This study is a prospective, observational, non-interventional cohort study to explore investigate the effects of neutrophil extracellular traps and damage-associated molecular pattern molecules on long term use of macrolides in adults with chronic respiratory disease.The study subjects were adult patients with chronic respiratory disease who met the inclusion criteria in the outpatient department from August 2021 to August 2023. A face-to-face questionnaire survey was conducted. ACT score was used for asthma control evaluation. Baseline data such as pulmonary function, FeNO, blood routine, induced sputum cell count, etc. were obtained. The use of hormones and other drugs was recorded. Inflammatory biomarkers were detected. 20ml venous blood was drawn to extract neutrophils to detect the expression of neutrophil extracellular traps and RT-PCR and ELISA were used to detect the expression of DAMPs. The total study duration was 2 years, with telephone visits every 3 months to assess chronic respiratory disease control and record subject compliance, unscheduled outpatient, emergency, and inpatient status.

ELIGIBILITY:
Inclusion Criteria:

* 1）Age ≥ 18 years; 2）Gender: not limited; 3）Diagnosis of asthma according to GINA guidelines (version 2021). 4）COPD was diagnosed according to GOLD guidelines (version 2021). 5）ACOS was diagnosed according to the consensus criteria for asthma-chronic obstructive pulmonary overlap syndrome (version 2021).

Exclusion Criteria:

* 1) Acute heart failure, severe organ failure, malignant tumors; 2) Other lung diseases such as pulmonary infection，pulmonary hypertension,tumor which seriously affect lung function, sputum cell classifi cation and other test results; 3) Pregnancy and lactation; 4) Recent surgery history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults With Chronic Respiratory Disease.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neutrophil Extracellular Traps and Damage-associated Molecular Pattern Molecules in 2 Years | baseline and 2years
  Using elisa to measure e-DNA and HMGB-1 concentrations in sputum from patients.
  Change=(Baseline concentrations -2 Years concentrations )

CONTACTS AND LOCATIONS:
Overall Officials: Haijin Zhao, M.D, Study Chair — Laboratory of Chronic Airway Diseases，NanfangH.
Locations (1):
- Haijin Zhao, Guangzhou, Guangdong, China